CLINICAL TRIAL: NCT07100626
Title: In Situ Clinical Trial Investigating the Ability of BlueCheck to Detect and Monitor Active Carious Lesions and Their Remineralization
Brief Title: In-situ Clinical Trial Assessing Ability to Detect and Monitor Active Caries and Their Remineralization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Incisive Technologies Pty Ltd (Industry)
Collaborators: Oral Health Research Institute, Indiana University School of Dentistry (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 25-I-126
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: BlueCheck — Caries Detection and Monitoring

SUMMARY:
The goal of this clinical trial is to evaluate whether BlueCheck® can accurately detect and monitor early-stage dental caries (tooth decay) and their remineralization in adults. Participants will wear partial dentures with partially demineralized human enamel specimens. The main questions it aims to answer are:

* Can BlueCheck® reliably detect early carious lesions with high sensitivity and specificity?
* Does BlueCheck® visually reflect changes in remineralized enamel lesions?

BlueCheck® results will be compared against standard diagnostic methods (e.g., Nyvad criteria, Diagnodent readings, surface microhardness) to see if BlueCheck® provides an objective, accurate, and visual method of detecting and monitoring early-stage caries.

Participants will:

* Wear a modified lower partial denture with four mounted enamel specimens for 28 days.
* Use only the study-provided fluoride containing toothpaste
* Attend weekly clinic visits for removal and laboratory analysis of one enamel specimen per week.
* Undergo regular oral health checks and provide diary entries tracking brushing and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* provide voluntary, written informed consent;
* be between 18 and 85 years old;
* understand and be willing, able and likely to comply with all study procedures and restrictions;
* be wearing a removable mandibular partial denture with sufficient room to accommodate four (4) human enamel specimens (4 mm round) in their partial denture on both sides (two specimens on each side, bilateral partial denture) or one side (4 specimens on one side, unilateral partial denture)
* be willing and capable of wearing their removable partial denture 24 hours a day for four (4), one-week treatment periods, maximum total duration four (4) weeks;
* be willing to allow study personnel to drill specimen sites in the posterior section of one or both sides of their lower partial denture (teeth and/or buccal flange area below the teeth); and
* be in good medical and dental health with no active caries or periodontal disease.
* have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/min; gum base stimulated whole saliva flow rate ≥ 0.8 mL/min).

Exclusion Criteria:

* currently be pregnant (self-reported), intending to become pregnant during the study period or breast feeding;
* currently have any medical condition that could be expected to interfere with the subject's safety during the study period;
* currently be taking antibiotics or have taken antibiotics in the two weeks prior to the beginning treatment;
* known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients;
* have participated in another clinical study or receipt of an investigational drug within 30 days of beginning treatment; or
* be taking fluoride supplements, required to use a fluoride mouthrinse or have received a professional fluoride treatment in the two weeks preceding specimen placement.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of BlueCheck to detect early stage carious lesions | Day 0
  BlueCheck will be applied to the early stage enamel carious lesions and visually assessed whether they are highlighted blue
Specificity of BlueCheck to not visual highlight sound enamel | Day 0
  BlueCheck will be applied to sound enamel samples and visually assessed whether they are highlighted blue.

SECONDARY OUTCOMES:
Change in BlueCheck colouration of remineralised artificial carious lesions | Day 1, 7, 14, 21 and 28
  Artificial carious lesions will be remineralised by application of fluoride containing toothpaste. Change in colouration of the lesions before and after remineralization in-situ will be compared to changes in surface microhardness over the same period.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lippert, PhD, Principal Investigator — Oral Health Research Institute, Indiana University School of Dentistry
Locations (1):
- Oral Health Research Institute, Indianapolis, Indiana, United States